CLINICAL TRIAL: NCT06641011
Title: The Effect of Rinsing Off or Blot-drying Silver Fluoride on the Retention of Subsequently-applied Resin- and Glass Ionomer-based Fissure Sealants in Permanent Molars Affected by Molar-Incisor Hypomineralization.
Brief Title: This Study Aims to Evaluate the Effect of Rinsing Off or Blot-drying Silver Fluoride on the Retention of Subsequently-applied Resin- and Glass Ionomer-based Fissure Sealants in Permanent Molars Affected by Molar-Incisor Hypomineralization.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Ballikaya, Associated Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TDH-2024-21181; TDH-2024-21181 (Other Grant/Funding Number: Hacettepe University Scientific Research Projects)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Molar Incisor Hypomineralisation; Children; Dental Caries
Keywords: Molar Incisor Hypomineralisation; Children; Silver Fluoride; Fissure Sealant; Glass ionomer; Silver-modified atraumatic restorative treatment
MeSH Terms: conditions — Molar Hypomineralization; Dental Caries

STUDY DESIGN:
Intervention Model Description: Randomization of molar teeth into six groups according to the restoration time, dental restorative material type, and conditions:
  Group 1: Restoration one week after silver fluoride application (n=72) Subgroup 1: Resin-based fissure sealant (n=36) Subgroup 2: Glass ionomer-based fissure sealant (n=36) Group 2: Immediate restoration after silver fluoride application (n=144) Subgroup 1: Blot-drying silver fluoride with cotton pellet followed by resin-based fissure sealant (n=36) Subgroup 2: Blot-drying silver fluoride with cotton pellet followed by glass ionomer-based fissure sealant (n=36) Subgroup 3: Rinsing silver fluoride off and air-drying of fissures followed by resin-based fissure sealant (n=36) Subgroup 4: Rinsing silver fluoride off and blot-drying of fissures followed by glass ionomer-based fissure sealant (n=36)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Resin based fissure sealant restoration one week after silver fluoride (AgF) application (Active Comparator): Resin-based fissure sealant restoration one week after silver fluoride (AgF) application
  Interventions: Device: Resin based fissure sealant restoration one week after silver fluoride (AgF) application
- Immediate resin based fissure sealant after blot drying silver fluoride (AgF) application (Active Comparator): Immediate resin based fissure sealant after blot drying silver fluoride (AgF) application
  Interventions: Device: Immediate restoration (resin- based) after blot-drying silver fluoride application
- Immediate GI-based fissure sealant after rinsing silver fluoride application (Active Comparator): Immediate GI-based fissure sealant after rinsing silver fluoride application
  Interventions: Device: Immediate restoration (GIC) after rinsing silver fluoride application
- Immediate GI-based fissure sealant after blot-drying of silver fluoride application (Active Comparator): Immediate GI-based fissure sealant after blot-drying of silver fluoride application
  Interventions: Device: Immediate restoration (GI- based) after blot-drying silver fluoride application
- Immediate resin-based fissure sealant after rinsing of silver fluoride application (Active Comparator): Immediate resin-based fissure sealant after rinsing of silver fluoride application
  Interventions: Device: Immediate restoration (Resin based) after rinsing silver fluoride application
- GI-based fissure sealant restoration one week after silver fluoride (AgF) application (Active Comparator): GI-based fissure sealant restoration one week after silver fluoride (AgF) application
  Interventions: Device: GI- based fissure sealant restoration one week after silver fluoride (AgF) application

INTERVENTIONS:
Device: Immediate restoration (resin- based) after blot-drying silver fluoride application — Blot-drying silver fluoride with cotton pellet followed by resin-based fissure sealant
  Other Names: Silver fluoride + glass ionomer sealant; Silver fluoride+ resin-based sealant
  Arms: Immediate resin based fissure sealant after blot drying silver fluoride (AgF) application
Device: Immediate restoration (GI- based) after blot-drying silver fluoride application — Blot-drying silver fluoride with cotton pellet followed by glass ionomer-based fissure sealant
  Arms: Immediate GI-based fissure sealant after blot-drying of silver fluoride application
Device: Immediate restoration (Resin based) after rinsing silver fluoride application — Rinsing silver fluoride off followed by resin-based fissure sealant
  Arms: Immediate resin-based fissure sealant after rinsing of silver fluoride application
Device: Immediate restoration (GIC) after rinsing silver fluoride application — Rinsing silver fluoride off and blot-drying of fissures followed by glass ionomer-based fissure sealant
  Arms: Immediate GI-based fissure sealant after rinsing silver fluoride application
Device: Resin based fissure sealant restoration one week after silver fluoride (AgF) application — Resin based fissure sealant restoration one week after silver fluoride (AgF) application
  Arms: Resin based fissure sealant restoration one week after silver fluoride (AgF) application
Device: GI- based fissure sealant restoration one week after silver fluoride (AgF) application — GI- based fissure sealant restoration one week after silver fluoride (AgF) application
  Arms: GI-based fissure sealant restoration one week after silver fluoride (AgF) application

SUMMARY:
The aim of this study is three-fold: 1. To evaluate the clinical performance of glass ionomer fissure sealants and resin fissure sealants when placed immediately after or one week following the application of silver fluoride on permanent molars affected by Molar-Incisor Hypomineralization in high caries-risk children. 2. To compare the effects of rinsing off the silver fluoride or not rinsing it off (blot-drying with cotton pellet) on sealant retention when the sealant is placed immediately after silver fluoride application, and 3. To measure the desensitizing effect of fissure sealant application following silver fluoride treatment on hypersensitive MIH molars.

DETAILED DESCRIPTION:
Teeth will be randomized in a parallel design based on the application of restoration time (immediate or one week later), sealant material type (resin or glass ionomer), and for immediate applications, the condition of silver fluoride before restoration (dried with cotton or rinsed gently). A total of 216 permanent molars will be included in the study.

Randomization of molar teeth into six groups according to the restoration time, dental restorative material type, and conditions:

ELIGIBILITY:
Inclusion Criteria:

* Patients and their parents who consent to participate and have signed the informed consent form.
* Patients with at least one permanent molar diagnosed with molar incisor hypomineralization based on EAPD guidelines.
* Fully erupted teeth with ICDAS I or II lesions that necessitate the application of fissure sealants.
* Teeth displaying demarcated opacities on the occlusal surface and at least one additional surface.

Exclusion Criteria:

* Teeth that have existing restorations or cavities.
* Patients currently receiving orthodontic treatment.
* Patients who are uncooperative during dental procedures.
* Teeth affected by dental fluorosis or enamel defects associated with specific syndromes.
* Children with systemic conditions requiring ongoing medication.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Retention Rate of Fissure Sealants with regard to the type of sealant and AgF pretreatment applied. | From enrollment to the end of treatment: 14 months (from July 2023 to October 2024). The first-year outcomes are planned for October 2025, and the second-year outcomes are planned for October 2026.
  The US Public Health Service criteria (secondary caries, anatomical form, marginal adaptation, marginal discoloration) will be used for clinical evaluation of restorations. The restorations will be evaluated at baseline and 1., 6., 12., 18., 24. months. Intra-oral photos will be taken directly after treatment and at control appointments to evaluate discoloration and seconder caries under magnification.

SECONDARY OUTCOMES:
Incidence of Caries | From enrollment to the end of treatment: 14 months (from July 2023 to October 2024). The first-year outcomes are planned for October 2025, and the second-year outcomes are planned for October 2026.
  The US Public Health Service criteria (secondary caries, anatomical form, marginal adaptation, marginal discoloration) will be used for clinical evaluation of restorations. The restorations will be evaluated at baseline and 1., 6., 12., 18., 24. months
Marginal Integrity of Sealants | From enrollment to the end of treatment: 14 months (from July 2023 to October 2024). The first-year outcomes are planned for October 2025, and the second-year outcomes are planned for October 2026.
  The US Public Health Service criteria (secondary caries, anatomical form, marginal adaptation, marginal discoloration) will be used for clinical evaluation of restorations. The restorations will be evaluated at baseline and 1., 6., 12., 18., 24. months
Tooth Sensitivity | From enrollment to the end of treatment: 14 months (from July 2023 to October 2024). The first-year outcomes are planned for October 2025, and the second-year outcomes are planned for October 2026.
  The Schiff Cold Air Sensitivity Scale (SCASS) will be used at 1, 6, 12, 18 and 24 months follow-ups to assess the presence of hypersensitivity in affected teeth by applying an air blast perpendicularly on the occlusal surface of the tooth for 1 second at a distance of 1 cm.
  The patient's response will be recorded according to the following scores:
  0 = subject does not respond to the stimulus;
  1. = subject does not respond to the stimulus but considers the stimulus to be painful;
  2. = subject responds to the air stimulus and moves away from the stimulus; and 3 = subject responds to the air stimulus, moves away from the stimulus, and requests an immediate cessation of the stimulus
Color and esthetic Changes | From enrollment to the end of treatment: 14 months (from July 2023 to October 2024). The first-year outcomes are planned for October 2025, and the second-year outcomes are planned for October 2026.
  Discoloration of the restorations will be recorded at 1, 6, 12, 18, and 24 months follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Ballikaya, DDS, PhD, Principal Investigator — Hacettepe University; Zafer Cehreli, DDS, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Dentistry, Department of Pediatric Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD is available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD is available from the corresponding author on reasonable request after October 2025
Access Criteria: IPD is available from the corresponding author on reasonable request.

REFERENCES:
- See also: Related Info — https://link.springer.com/article/10.1007/s00784-021-04236-5